CLINICAL TRIAL: NCT05066334
Title: Intervertebral Disc Regeneration Mediated by Autologous Mesenchymal Stem/Stromal Cells Intradiscal Injection: a Phase IIB Randomized Clinical Trial - DREAM Trial
Brief Title: Efficacy of Intradiscal Injection of Autologous BM-MSC in Subjects With Chronic LBP Due to Multilevel Lumbar IDD
Acronym: DREAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Center for Outcomes Research and Clinical Epidemiology, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DREAM (GR - 2018-12367168); 2019-002749-40 (EudraCT Number)
Record Dates: First submitted 2021-07-27; First posted 2021-10-04 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-08

CONDITIONS: Intervertebral Disc Degeneration; Chronic Low-back Pain
Keywords: Low Back Pain; Spine; Intervertebral Disc Degeneration; Mesenchymal Stem Cells; Bone Marrow
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — Therapeutics; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in 2 arms of 26 patients and followed up for 24 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The randomization will be centralized and stratified on the investigation center. Treatment allocation will be performed 24 hour-a-day online by a central randomization web-service. The patient identification must be unique within all randomizations performed. For double-blind trial the randomization result will be a treatment code. Blinding or masking will be carried out at all stages of packaging and conditioning for shipping following the treatment allocation. Injections used for all groups will be clear and indistinguishable from each other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Arm (Experimental): Two procedures:
  1. Bone marrow harvesting from the posterior superior iliac crest region
  2. Single injections of a dose of 15 million of autologous BM-MSC for each disc affected by IDD (up to 3 discs) via imaging control
  Interventions: Drug: Autologous BM-MSC
- Sham Procedure (Sham Comparator): Two sham procedures:
  1. Simulated bone marrow harvesting without insertion into the posterior iliac crest region
  2. Simulated injection under only local anaesthesia without disc injection and without placebo injection.
  Interventions: Procedure: Sham

INTERVENTIONS:
Drug: Autologous BM-MSC — intradiscal injection of autologous bone marrow mesenchymal stromal cells
  Other Names: Treated
  Arms: Active Arm
Procedure: Sham — local anaesthesia, no disc injection, no placebo injection
  Other Names: Untreated
  Arms: Sham Procedure

SUMMARY:
DREAM is a phase II B efficacy monocentric, prospective, randomized, controlled double blinded trial, comparing intra-discal autologous adult bone marrow mesenchymal stem cells (BM-MSC) therapy and sham treated controls in subjects with chronic (> 6 months) Low Back Pain (LBP) due to lumbar multilevel (max. 3 levels) intervertebral disc degeneration (IDD) unresponsive to conventional therapy.

Duration of the recruitment period has been estimated to be 12 months. The efficacy of intradiscal injection of autologous BM-MSC in reducing chronic LBP due to multilevel lumbar IDD will be evaluated after 24 months in terms of pain relief (VAS), functionality (ODI) and quality of life (SF36).

DETAILED DESCRIPTION:
Low back pain (LBP) is the global leading cause of disability, and furthermore rates sixth in terms of overall disease burden, in both developed and developing countries. LPB is a condition of all ages, from children to elderly, affecting 60-70 percent of the global population during life, and ~700 million people each year. LBP prevalence increases with age, and with populations ageing worldwide, the societal and economic burden associated with LBP will increase substantially over coming years.

Current LBP therapies are aimed at pain reduction, and do not provide restorative treatment. Such conservative strategies (e.g. painkillers and musculoskeletal rearrangement by manual and physiotherapy) rarely address the actual cause of LBP.

In a healthy spine, intervertebral discs (IVDs) separate the vertebrae to provide complex spinal flexibility while supporting large spinal loads. Intervertebral disc degeneration (IDD) is widely recognized as a major contributor to LBP, responsible for at least 40 percent of LBP cases. A key characteristic of IVD degeneration is loss of matrix integrity, thereby causing biomechanical functional failure.

Today, no therapy can restore IVD function or provide long-term relief from symptomatic IDD. New treatment strategies concentrate on treating IDD at an early stage. Stem cell research offers exciting possibilities, and advanced cell-based therapies are considered highly promising strategies in treating IVD degeneration and LBP. Encouraging results suggest that cell-based, regenerative therapies may provide the world first effective therapy for this common and debilitating disease.

The objective of DREAM is to generate efficacy and tolerability profiles of a single injection of 15 million of cells/ml of autologous BM-MSC for each disc affected by IDD (up to 3 discs) versus sham procedure. The potential of BM-MSC to lead to a disease-modifying therapeutic option for the treatment of this chronic and debilitating disease will be assessed by Magnetic Resonance Imaging (MRI) after 6 months, 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Symptomatic chronic LBP due to moderate IDD (modified Pfirrmann score 3-4, Griffith score 3-7) at max.3 levels of the lumbar spine unresponsive to conservative treatment, physical and medical for at least 6 months. Physical treatment includes physiotherapy. Medical treatments includes nonsteroidal anti-inflammatory drugs (NSAID), paracetamol, opioids and myorelaxant.
* Annulus fibrosus intact, demonstrated by MRI.
* Pain baseline > 40 mm on VAS (0- 100).
* NSAID washout of at least 2 days before screening.
* Painkillers washout of at least 24 hours before screening.
* For females of childbearing potential, a negative pregnancy test must be documented at Screening.
* Men and women should use effective contraception during treatment and for at least 24 months after BM-MSC discontinuation. As a precautionary measure, breast-feeding should be discontinued during treatment with BM-MSC and should not be restarted after discontinuation of BM-MSC.

Exclusion Criteria:

* Congenital or acquired diseases leading to spine deformations that may upset cell application (scoliosis, isthmus lesion, sacralization and hemisacralization, degenerative spondylolisthesis).
* Spinal segmental instability assessed by dynamic X-Ray.
* Symptomatic facet joints syndrome on MRI (facet joints hyperintensity and hypertrophy evaluated at coronal T2 weighted MRI).
* Prior to the screening visit, has received:
* Oral corticosteroid therapy within the previous 3 months, OR
* Intramuscular, intravenous or epidural corticosteroid therapy within the previous 3 months
* Presence of a 4th level with symptomatic IDD (modified Pfirrmann score 3-4, Griffith score 3-7) in the lumbar spine.
* Spinal canal stenosis (Schizas score > B).
* History of spinal infection.
* Lumbar disc herniation and sciatica.
* Endplate abnormality such as Schmorl's Nodes.
* Previous discal puncture or previous spine surgery.
* IDD with Modic II and III changes on MRI images.
* Patients not eligible to the intravertebral disc surgery.
* Patients who have the risk to undergo a surgery in the next 6 months.
* Patients with local infusion device/devices for corticosteroids.
* Obesity with body mass index (BMI in Kg/size in m^2) greater than 35 (obesity grade II).
* Participation in another clinical trial or treatment with another investigational product within 30 days prior to inclusion in the study.
* Abnormal blood tests: hepatic (alanine amino transferase [ALT] and/or aspartate aminotransferase [AST] > 1.5 × upper limit of normal [ULN]), renal, pancreatic or biliary disease, blood coagulation disorders, anemia or platelet count of < 100 × 10^9/L.
* Pregnant or lactating women, or premenopausal women not using an acceptable form of birth control, are ineligible for inclusion. Contraception will be maintained during treatment and until the end of relevant systemic exposure. Additional pregnancy testing will be performed at the end of relevant systemic exposure. The patients will be required to use contraception from initial treatment administration until 24 months after the last dose of study drug.
* In each case of delayed menstrual period (over one month between menstruations) confirmation of absence of pregnancy is strongly recommended.
* Positive serology for following infection: Syphilis, HIV, Hepatitis B, or C.
* Contraindication to MRI assessed by the investigator.
* Intolerance or allergy to local anaesthesia.
* Any history of Cancer or immunodeficiency disease.
* Previous transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain Change | From Baseline to Month 24
  Changes in pain will be evaluated on Visual Analogic Scale (VAS) between baseline and month 24. VAS scale ranges from 0 to 100, where 0 represents no pain and 100 represents the worst pain imaginable.
Functional disability index evaluation | From Baseline to Month 24
  Functional disability changes will be assessed on Oswestry Disability Index (ODI, also known as the Oswestry Low Back Pain Disability Questionnaire) at month 24 compared with baseline. ODI scale ranges from 0 to 50 and allows evaluation of disability (0 - 20 percent: minimal disability; 20 - 40 percent: moderate disability; 40 - 60 percent: severe disability; 60 - 80 percent: crippled; 80 - 100 percent: bed-bound or exaggerating their symptoms).

SECONDARY OUTCOMES:
Disability evolution | Baseline, 3, 6, 12 and 24 months
  Disability evolution includes Short Form-36 Health Survey (SF-36) scores. SF-36 scores consist of eight 0-100 scaled scores (vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning and mental health) where a lower score corresponds to more disability and a higher score corresponds to less disability.
Quality of life evolution | Baseline, 3, 6, 12 and 24 months
  Quality of life evolution includes global assessment by the patient and the physician.
  The global assessment by the patient and the physician involves evaluation of: - Overall pain intensity in the lumbar spine (1 = none, 2 = mild, 3 = moderate, 4 = severe, 5 = extreme); - patient's global assessment of disease activity (1 = very good, 2 = good, 3 = fair, 4 = poor, 5 = very poor); - physician's global assessment of disease activity (1 = very good, 2 = good, 3 = fair, 4 = poor, 5 = very poor).
Drug consumption of rescue painkillers medication | Baseline, 3, 6, 12 and 24 months
  The decrease/increase in the use of rescue medication will be recorded throughout the study duration by a diary file. A reduction in dose or frequency of administration of painkillers is an indirect marker of the benefits of MSC therapy.
Measurement of pain | Baseline, 3, 6, 12 and 24 months
  Assessed by Visual Analogic Scale (VAS). VAS pain scale ranges from 0 to 100: where 0 represents no pain and 100 represents the worst pain imaginable. In brief, the patients will fill VAS tests indicating the amount of pain experienced at rest and in motion.
Employment and work status assessment | Baseline and 24 months
  For this the investigators will assign each of the patients to one of 4 categories designated as "employable" which included those who were unemployed due to pain, employed but on sick leave, laid off, or working. The other categories include retired, disabled, and elderly at least 60 years of age, eligible for social security.
Structural assessment | Baseline, 6, 12 and 24 months
  Evolution of affected disc(s) by quantitative Magnetic Resonance Imaging (MRI) density measurements in T2 and T1 spin/echo and T1 rho weighted images used as an indication of disc fluid and glycosaminoglycans (GAG) content. The "quality" of the patient's lumbar disc/discs will be monitored non invasively using T2 weighted MRI sagittal images and, in T1 spin/echo MRI. Lumbar disc grading will be performed in the sagittal T2 weighted images by two physicians independently who were experienced in MRI of the spine. They will review each intervertebral disc from L1-2 to L5-S1 by the modified Pfirrmann criteria. The modified Pfirrmann grading system assesses degenerated intervertebral discs by MRI for the asymmetry in disc structure, distinction of the nucleus and the annulus, signal intensity of intervertebral discs and height of intervertebral discs and assigns grade 1 to 8 for disc degeneration.
Evaluation of costs | 12 and 24 months
  The investigators will compare the medical and non-medical costs between the two groups of patient. For this purpose, resource use in each arm will be collected in physical units in the eCRF (electronic case report form) at the clinical centre as follows:
  * Acute care medical hospitalisations related to IDD
  * Acute care surgical hospitalisations related to IDD
  * Rehabilitation hospitalisations related to IDD
  * Analgesics
  * Work disruption
Body Mass Index evaluation | Baseline, 3, 6, 12 and 24 months
  Evaluation of changes in Body Mass Index (BMI) through the measurement of weight (kg) and height (m) of each subject enrolled in the study.
Haematological evaluation: safety parameter | Baseline, 3, 6, 12 and 24 months
  The investigators will assess the percentage of patients who will develop haematological disorders. For this reason, participants will undergo blood sampling for routine laboratory testing to determine haematological parameters (haematocrit, haemoglobin, RBC, WBC) to monitor the physiological status of the patient.
Coagulation status: safety parameter | Baseline, 3, 6, 12 and 24 months
  The investigators will assess the incidence of disorders related to coagulation. For this reason, participants will undergo blood sampling for routine laboratory testing to determine coagulation parameters (INR, PTT) to monitor the coagulation status and hemostasis risks of each subject.
Metabolic functions: safety parameter | Baseline, 3, 6, 12 and 24 months
  The investigators will evaluate the incidence of metabolic alteration in patients recruited. For this reason, participants will undergo blood sampling for routine laboratory testing to determine biochemical parameters (Electrolytes, Creatinine, ALT, AST, AP, Bilirubin) to monitor the metabolic function of liver and kidney.
Inflammation: safety parameter | Baseline, 3, 6, 12 and 24 months
  Blood sampling will be used to determine the concentration of C-Reactive Protein (CRP). Participants will undergo blood sampling for routine laboratory testing to monitor inflammatory response in each subject.
Urinalysis | Baseline, 3, 6, 12 and 24 months
  Participants will undergo to urinalysis which consists in routine urine tests for the semiquantitative assessment of urinary characteristics to monitor the physiological status of the subjects.
Spine examination | Baseline, 3, 6, 12 and 24 months
  Participants will undergo to spine examination for the identification of relevant clinical signs. The clinicians will evaluate: abnormalities in gait (pattern of walking); spinal range of motion (eg, bend forward); posture and spinal alignment (such as scoliosis or kyphosis).
Specific Adverse Events Evaluation | Baseline, 3, 6, 12 and 24 months
  Participants will be interviewed by the investigator to fill a study-specific Adverse Events checklist for recording of symptoms and complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Vadalà, MD, PhD, Principal Investigator — Campus Bio-Medico University of Rome
Locations (1):
- Campus Bio-Medico University of Rome, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No